CLINICAL TRIAL: NCT03433404
Title: Soft Tissue Mobilization for Lumbopelvic Pain in the Third Trimester of Pregnancy
Acronym: STM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: L17-191
Record Dates: First submitted 2018-01-29; First posted 2018-02-14 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain; Pregnancy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft Tissue Mobilization (Experimental): The arm will utilize a Physical Therapy technique call soft tissue mobilization.
  Interventions: Procedure: Soft Tissue Mobilization
- Soft Tissue Massage (Active Comparator): This arm will utilize standard soft tissue massage applied to the low back in pregnant patients complaining of third trimester low back pain.
  Interventions: Procedure: Soft Tissue Massage
- No manual treatment (No Intervention): Group will still receive acetaminophen, heating pad application, and/or rest which is standard of care.

INTERVENTIONS:
Procedure: Soft Tissue Mobilization — The technique has been described previously in other descriptions. However, the main goal of this treatment is to address the LDSIL in the manner described previously in order to mobilize the soft tissue in the area.
  Arms: Soft Tissue Mobilization
Procedure: Soft Tissue Massage — For sMass, the subject will be positioned on her side opposite to the most painful side of the lumbosacral spine with the hips flexed to 45 degrees and knees flexed to 90 degrees (with a pillow positioned between them). The investigator will perform superficial (light stroke) massage to the painful side of the lumbosacral region for 5 minutes
  Arms: Soft Tissue Massage

SUMMARY:
Back pain is one of the most common complaints in pregnancy. It is caused by the growing pregnant abdomen which then strains the lower back and pelvis. Often Obstetricians recommend rest, Tylenol, pelvic support belts, or exercise. Typically, these do not provide the patient much relief. A physical therapy treatment known as soft tissue mobilization (tSTM) has been shown to be helpful in treating various types of pain. This study will explore whether tSTM can improve back pain in pregnancy.

DETAILED DESCRIPTION:
Context: Lumbopelvic pain is one of the most common complaints in pregnancy, as increasing hormone levels cause joint laxity and the gravid uterus weakens abdominal muscles and increases lumbar muscle strain. Obstetricians often recommend rest, exercise, heating pad application, acetaminophen, or pelvic support belts. Patients often complain of minimal relief from these recommendations. Many experience recurrent lumbopelvic pain in a subsequent pregnancy. Additionally, lumbopelvic pain can contribute to disability and sick leave during the pregnancy. This is the first study to investigate whether soft tissue mobilization improves lumbopelvic pain in the third trimester.

Objective: To investigate whether a physical therapy intervention known as transverse friction massage or soft tissue mobilization improves third trimester pregnancy related lumbopelvic pain.

Design: Randomized pre-test and post-test comparison group design. Setting: Texas Tech University Health Sciences Center, Center for Rehabilitation Research, Lubbock, TX, USA.

Participants: 48 subjects between the 18-45 years of age with a singleton gestation in the third trimester with pregnancy related lumbopelvic pain.

Methods: Subjects consented for the study will be diagnosed by the Obstetrician with PRLPP by clinical tests, including the posterior pelvic pain provocation test, active straight leg raise test, and the long dorsal sacroiliac ligament test. Subjects will be randomized to one of three groups: no manual treatment (noManRx), superficial massage (sMass), and soft tissue mobilization (tSTM). All groups will receive standard care, which includes acetaminophen, heating pad application, and/or rest. Subjective questionnaires including the numeric pain rating scale (NPRS), the Oswestry Disability Index (ODI), and the Global Rating of Change (GROC) will be administered for baseline prior to allocated intervention. The Pressure Pain Threshold (PPT) will be measured via algometry. Those receiving sMass and tSTM will receive prescribed standard care as well as sMass or tSTM every 1-2 weeks by an investigator as well as daily sMass or tSTM at home.

Main outcome measures: (1) Pain using NPRS, (2) disability using ODI, (3) overall change in pain pre- and post-treatment using GROC, (4) pressure pain threshold via algometry.

Expected results: It is anticipated that this soft tissue mobilization technique known as transverse friction massage will decrease lumbopelvic pain in the third trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Subjects 18-45 years old
* singleton gestation in the third trimester (28 weeks and on)
* pregnancy-related lumbopelvic pain
* capable of following basic instructions.

Exclusion Criteria:

* Subjects with a history of lumbopelvic pain that required healthcare management within a year prior to pregnancy
* acute infectious or inflammatory process
* diagnosed mental health disorder
* substance abuse
* documented diagnosis of fibromyalgia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Inclusion Criteria: (1) Subjects 18-45 years old with (2) singleton gestation in the third trimester (28 weeks and on); (3) pregnancy-related lumbopelvic pain; and (4) capable of following basic instructions.
  Exclusion Criteria: (1) Subjects with a history of lumbopelvic pain that required healthcare management within a year prior to pregnancy, (2) acute infectious or inflammatory process, (3) diagnosed mental health disorder; (4) substance abuse; (5) documented diagnosis of fibromyalgia.
Enrollment: 26 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Pain using NPRS (Numerical Pain Rating Scale) | through study completion, an average of 1 year
  The NPRS is a scale from 0 to 10 that is commonly used to measure intensity of pain, with 0 representing no pain and 10 representing extreme pain. It is easy to understand and complete that is also valid and reliable. Due to the nature of fluctuating intensity of pain, subjects will use a NPRS to log their current pain, least pain, and most pain each day at home and at the obstetric clinic before the respective treatment. The daily pain score will be averaged, then averaged across each week. The NPRS scores will be also be used to evaluate the change between the overall pain level at the beginning and end of subject's participation. The aim throughout the study is to see a reduction in the overall numerical pain scale rating. For example, if a patient comes in with a pain scale rating of 10, the hope is that after a series of treatments, the pain scale will go down to indicate an improvement in overall pain.
disability using ODI (Oswestry Disability Index) | through study completion, an average of 1 year
  Back pain and its effect on disability can be evaluated using the ODI. It is a brief 10 question survey on the effect of back pain on daily activities, such as personal care, walking, lifting, sitting, standing, sex life, social life, traveling. Each answer in each section is scored 0 to 5, 0 if the first box is checked (0 if it causes no disability) and 5 (maximal disability) if the last box is checked. The final score is expressed as a percentage out of a total score of 50. It is usually used for lumbar back pain, but has been shown to be specifically valid for sacroiliac joint pain. The ODI questionnaire will be filled out by subjects at the initial session and at the end of the final treatment session.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No